CLINICAL TRIAL: NCT02183948
Title: Effect of Oxytocin on Masked Facial Expressions: an fMRI Study
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Keith Kendrick, Professor / Research group leader, University of Electronic Science and Technology of China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: UESTC-SCAN-01; UESTC-SCAN-01 (Other Grant/Funding Number: NSFC)
Record Dates: First submitted 2014-06-30; First posted 2014-07-08 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-03

CONDITIONS: Facial Expressions
Keywords: treatment; mask face exoressions; genier
MeSH Terms: conditions — Facial Expression | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- oxytocin (Experimental): nasal spray
  Interventions: Drug: Oxytocin
- Placebo (Placebo Comparator): nasal spray
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin
  Arms: oxytocin
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose is to test whether oxytocin has an effect on masked facial expressions

DETAILED DESCRIPTION:
The neuropeptide oxytocin (OXT) has been shown to modulate several aspects of human social cognition. Although the exact mechanisms behind these effects remain unclear, recent research suggests that OXT modulates the perception of cues that are important for interpersonal processing, particularly emotional facial expressions. Using a backward masking procedure and functional magnetic resonance imaging, we investigated the modulatory effects of intranasal OXT on the processing of sub-liminally presented emotional faces. In a double-blind placebo-controlled between-subject pharmaco-fMRI experiment healthy volunteers received either 24IU of intranasal oxytocin or placebo 45mins before they were presented emotional (happy, angry, fearful, sad, disgusting) faces and mirror-reversed neutral faces masked by neutral faces of the same individual. To ensure attentional processing of the faces subjects were required to perform a simple gender decision task in the scanner and a recognition memory task afterwards. All subjects were additionally assessed for their state and trait anxiety and depression as well as empathy. For the analysis, we will use matlab, SPM and SPSS to conduct structural ROI analysis and two Sample t test.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects, no smoke or drink alcohol, coffee or other stimulants during the day before Experiment.

Exclusion Criteria:

* history of head injury; pregnancy; uterine cavity operations were took within one year; medical or psychiatric illness; rhinitis in case they may not fully absorb the spray.

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2014-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Number of participants with neuro activity to facial expressions | one week